CLINICAL TRIAL: NCT07305246
Title: Clinical Study of SHR-A1811 With or Without Letrozole in Neoadjuvant Therapy for Early-Stage HR-Positive, HER2-Low Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yingying Xu, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-122
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-A1811 Combined with Endocrine Therapy (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Letrozole
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- Standard Chemotherapy Group (Active Comparator)
  Interventions: Drug: TAC/AC-T

INTERVENTIONS:
Drug: SHR-A1811 — Intravenous infusion at 4.8 mg/kg per dose, administered once every 3 weeks (Q3W). Each 3-week (21-day) period constitutes one treatment cycle, totaling 8 cycles.
  Administration is via intravenous infusion. The initial infusion duration is 90±10 minutes (including the flush phase).
  If no infusion-related reactions occur after the first administration, subsequent infusions may be shortened to approximately 30 minutes (not less than 20 minutes, including the flush phase).
  Arms: SHR-A1811; SHR-A1811 Combined with Endocrine Therapy
Drug: Letrozole — 2.5 mg orally once daily, taken continuously.
  Arms: SHR-A1811 Combined with Endocrine Therapy
Drug: TAC/AC-T — Recommended standard dose
  Arms: Standard Chemotherapy Group

SUMMARY:
This is a prospective, randomized, multi-cohort, Phase II clinical trial. The study plans to enroll 120 patients with early-stage or locally advanced, HR-positive, HER2-low breast cancer. The primary objective is to evaluate the efficacy and safety of SHR-A1811 with or without endocrine therapy compared to standard chemotherapy as neoadjuvant treatment.

Eligible subjects will be randomized centrally via an Interactive Web Response System (IWRS) using a block randomization method. Participants will be assigned in a 1:1:1 ratio to one of three treatment cohorts:

Cohort A: SHR-A1811 plus endocrine therapy (letrozole ± ovarian function suppression [OFS]) Cohort B: SHR-A1811 monotherapy Cohort C: Standard chemotherapy (investigator's choice of A/EC-T or TEC regimen)

Neoadjuvant Treatment:

Subjects in Cohorts A and B will receive 8 cycles of their assigned regimen. Subjects in Cohort C will receive standard chemotherapy as per the chosen protocol.

Treatment will continue until completion of the regimen, occurrence of unacceptable toxicity, withdrawal of consent, or discontinuation at the investigator's discretion.

Assessments:

Tumor imaging for efficacy evaluation will be performed every 2 cycles, with responses assessed according to RECIST v1.1 criteria. Subjects who complete neoadjuvant treatment and are deemed eligible for surgery will undergo surgical intervention within 4 weeks after treatment completion. Pathological response will be assessed from the surgical specimen. Both radiological and pathological evaluations will be based on the assessments conducted at the study site.

Adjuvant Therapy:

Following surgery, all subjects will receive standard adjuvant endocrine therapy as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥18 years and ≤70 years;
2. Histopathologically confirmed invasive breast cancer with no prior systemic anticancer therapy for breast cancer;
3. Histopathologically confirmed HR-positive (ER ≥1% and/or PR ≥1%) with HER2-low expression (defined as IHC 1+/2+ and FISH negative);
4. Stage II-III breast cancer (cT2-cT4 or N+, cM0) according to the 8th edition AJCC Breast Cancer Staging Manual;
5. At least one measurable target lesion per RECIST V1.1;
6. ECOG performance status score of 0 to 1;
7. Organ function levels must meet the following requirements (no corrective therapy with blood components or growth factors within 14 days prior to first dose):

   1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥100×10^9/L, hemoglobin ≥ 90 g/L;
   2. Hepatic and renal function: Albumin level ≥ 3.0 g/dL, total bilirubin ≤ 1.5×upper limit of normal(ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN, alkaline phosphatase ≤ 2.5×ULN, blood urea nitrogen and serum creatinine ≤ 1.5×ULN or creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula);
   3. Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
   4. Echocardiogram (ECHO) showing left ventricular ejection fraction (LVEF) ≥ 50%;
   5. QTcF ≤ 470 msec;
8. Pregnancy tests must be performed within 7 days prior to treatment initiation for premenopausal women of childbearing potential. Serum pregnancy tests must be negative, and participants must not be breastfeeding. All enrolled patients must use adequate barrier contraception throughout the treatment cycle and for 6 months post-treatment;
9. Voluntary participation in the study, signed informed consent, good compliance, and willingness to attend follow-up visits and undergo study-related procedures.

Exclusion Criteria:

1. Breast cancer not confirmed by histopathological examination;
2. Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer;
3. Prior receipt of any form of antitumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
4. Concurrent administration of any other form of antitumor therapy;
5. History of other malignancies within the past 5 years, except for cured basal cell carcinoma of the skin and cervical carcinoma in situ;
6. Participation in other drug clinical trials within 4 weeks prior to randomization;
7. Administration of live or attenuated vaccines within 4 weeks prior to randomization;
8. Undergone major non-breast cancer-related surgical procedures within 4 weeks prior to randomization, or not yet fully recovered from such procedures;
9. Presence of any active autoimmune disease or history of autoimmune disease with potential for recurrence, including but not limited to: autoimmune hepatitis, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (subjects controllable solely with hormone replacement therapy may be included); subjects with skin conditions not requiring systemic treatment such as vitiligo, psoriasis, or alopecia; controlled type 1 diabetes managed with insulin therapy; or childhood asthma in complete remission requiring no intervention in adulthood may be included; subjects with asthma requiring medical intervention with bronchodilators;
10. History of immunodeficiency disorders, including HIV-positive status, other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
11. Uncontrolled or significant cardiovascular or cerebrovascular disease, including (but not limited to): occurrence of any of the following within 6 months prior to first dosing: congestive heart failure (NYHA Class III or IV), myocardial infarction or cerebral infarction (excluding lacunar infarction), pulmonary embolism, unstable angina, or presence of treatable arrhythmia at screening; Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, or unclassified cardiomyopathy); History of clinically significant QTc prolongation, second-degree type II atrioventricular block or third-degree atrioventricular block, or QTc interval (F method) >470 msec (females); atrial fibrillation (EHRA classification ≥2b); uncontrolled hypertension deemed unsuitable for study participation by the investigator;
12. Subjects with known or suspected interstitial pneumonia; other conditions within three months prior to first dosing that may interfere with interfering with drug-related pulmonary toxicity monitoring or management, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/obstructive bronchiolitis, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), obstructive/restrictive lung disease, or any autoimmune, connective tissue, or inflammatory disease affecting the lungs, such as rheumatoid arthritis, Sjögren's syndrome, or sarcoidosis, or prior history of total lung replacement;
13. Active hepatitis B (HBsAg positive and HBV DNA ≥ 500 IU/mL), hepatitis C (HCV antibody positive and HCV RNA above upper limit of normal range), or cirrhosis; or severe infections requiring antibiotics, antivirals, or antifungals for control;
14. Known hereditary or acquired bleeding or thrombotic tendencies (e.g., hemophilia, coagulation disorders, etc.);
15. Known allergy or contraindication to the study drug or its excipients;
16. Pregnant or lactating female patients; female patients of childbearing potential with a positive baseline pregnancy test; or female patients of childbearing potential unwilling to use effective contraception throughout the study period;
17. Concomitant conditions judged by the investigator to pose a serious threat to patient safety or interfere with study completion (including but not limited to uncontrolled severe hypertension, severe diabetes, active infections, etc.);
18. History of defined neurological or psychiatric disorders, including epilepsy or dementia, or any other condition deemed by the investigator to make the patient unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
tpCR：ypT0-is/ypN0 | From enrollment to the end of surgery

SECONDARY OUTCOMES:
ORR | From enrollment to the end of treatment，an average of 1 year
EFS | From enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.